CLINICAL TRIAL: NCT07071506
Title: New Methods for Evaluating Preventive Migraine Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UAarhus_Chronic migraine
Record Dates: First submitted 2025-05-28; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Migraine; Migraine With or Without Aura; Headache Disorders; Chronic Migraine, Headache
Keywords: Headache; Chronic migraine; Balanced placebo design; Treatment effects; Adverse events
MeSH Terms: conditions — Migraine Disorders; Headache Disorders; Headache

STUDY DESIGN:
Intervention Model Description: Double-blinded randomized controlled cross-over design where patients receive
  1) Fremanezumab or 2) placebo, twice.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Active Comparator): Active drug
  Interventions: Drug: Active drug for chronic migraine treatment.
- Placebo group (Placebo Comparator): Inactive placebo
  Interventions: Drug: Placebo Subcutaneous injection

INTERVENTIONS:
Drug: Active drug for chronic migraine treatment. — Standard dose of Fremanezumab, 225 mg (Ajovy) injected subcutaneously
  Arms: Active group
Drug: Placebo Subcutaneous injection — Inactive placebo (saline) injected subcutaneously in the same volume as the active drug
  Arms: Placebo group

SUMMARY:
The study aims to estimate treatment effects in a balanced placebo design (BPD) to specify to which extent contextual factors interact in preventive migraine treatment and influence adverse event occurrence in patients with chronic migraine. Using a clinical within-subjects design, patients with chronic migraine will receive four treatment conditions in a randomized order.

DETAILED DESCRIPTION:
The existing paradigm for testing the effect of treatment is the double-blind RCT comparing an active drug to an inactive placebo. This comparison is done in order to control for contextual and psychological factors such as the patients' treatment expectations - a key factor in placebo responses. However, recent studies have indicated that some assumptions underlying the RCT may be incorrect and may lower the assay sensitivity and miscalculate the actual drug response. The so-called balanced placebo design targets some of the shortcomings of the RCT by balancing the information given to the patients with the actual treatment administered. In this project, patients suffering from chronic migraine will receive a total of 4 injections over 8 months. Half of them are femanezumab, while the other half are placebo (an inactive injection). The injections (fremanezumab and placebo) look the same, and neither the patient nor the investigator know which injection will be administered. The order will be randomized. The injections are given with different information about what the patients are receiving. To avoid a carry-over effect, the patients will receive one injection every second month. The first month will be without treatment whereupon the patient will receive the first injection. During the first 28 days before and after each administration, patients rate outcome measures in an electronic pain/headache diary at home. In addition, they will also fill out questionnaires assessing their quality of life, psychological parameters and the headache burden.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (18-65 years)
2. ≥ 1-year history of migraine with or without aura according to the International Classification of Headache Disorders (ICHD-3) diagnostic criteria
3. Known chronic migraine (headache occurring ≥ 15 days per month for > 3 months, which on at least 8 days per month has the features of migraine headache) diagnosed before age 50
4. Qualifying for preventive migraine treatment (screened by neurologist)
5. Ability to speak and read Danish

Exclusion Criteria:

1. Use of onabotulinumtoxinA as preventive migraine treatment during the 4 months before screening
2. Use of other preventive migraine treatment other than CGRP antagonists (However, participants are allowed to be on one stable preventive medication (antidepressant, calcium channel blockers, beta blockers or antiepileptic)- 2 months prior to screening until end of study , if necessary), devices for migraine prevention such as transcranial magnetic stimulation and use of nerve blocks 3 months prior to screening
3. Use of opioid or barbiturate medications in the last four weeks before participation in the study
4. Secondary headache disorders including medication overuse headache
5. Severe psychiatric, vascular disease, or known liver disease
6. Alcohol abuse, drug abuse, or substance abuse
7. Current or planned pregnancy and lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Moderate/severe headache days | Through study completion, an average of 8 months
  Total number of moderate/severe headache days will be measured 28 days before and after each treatment administration. Headache days will be recorded by the presence of headache (yes/no), peak pain intensity (mild/moderate/severe), and duration (< 4h or ≥ 4h), acute medication intake type (triptan/ergotamine/other) and migraine associated symptoms.
Headache/pain intensity | 8 months
  Headache/pain intensity rated on a 11-point Numerical Rating Scale (0=no pain; 10=worst pain intensity) will also be measured 28 days before and after each treatment administration.
Adverse events | 24 hours, 14 and 28 days after each treatment administration
  Occurrence of adverse events in each treatment condition recorded by the presence of adverse events ascribed to the treatment, measured by free recall and by prompting.

SECONDARY OUTCOMES:
Migraine days | Through study completion, an average of 8 months
  Total number of migraine days will be measured 28 days before and after each treatment condition.
Intensity of migraine | Through study completion, an average of 8 months
  A categorical, four-point rating scale will be used to rate each migraine day as absent, mild, moderate, or severe. It is is graded mild when it does not inhibit work or other activities, moderate when it inhibits but does not prohibit work or other activities, and severe when it prohibits work and other activities.
Acute treatment utilization | Through study completion, an average of 8 months
  The use of acute migraine medication will be recorded, including the number of days and the specific drug used.
Positive and negative affect (PANAS) | Pre-treatment and 28 days after each treatment administration
  PANAS will be used to measure positive and negative emotions or feelings pre- and post-treatment of each treatment condition. Positive affectivity refers to positive emotions and expressions. Negative affectivity, on the other hand, refers to negative emotions and expressions. This scale consists of words that describe different emotions and is scored on a Likert scale ranging from 1 to 5 (1= Very slightly or Not at all, 2=little, 3=moderately, 4=quite a bit and 5 =extremely).
Hospital Anxiety and Depression Scale (HADS) | Pre-treatment and 28 days after each treatment administration
  It is a 14-item measure designed to assess anxiety and depression symptoms. It is rated on a 4-point Likert scale. It will be measured pre- and post-treatment of each treatment condition.
Quality of life (SF-12) | Pre-treatment and 28 days after each treatment administration
  Short-form-12 (SF-12) is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It consists of two components- physical (PCS-12) and mental (MCS-12). The summary scores are scored using norm-based scoring, where means of 50 and standard deviations of 10 are achieved.
HIT-6 | Pre-treatment and 28 days after each treatment administration
  Headache impact test (HIT-6) measures the impact that headache has on social functioning, role functioning, vitality, cognitive functioning, and psychological distress. It consists of 6 questions. Each question can be answered with 5 responses (never, rarely, sometimes, very often, or always), which has the following numerical values (6, 8, 10, 11, and 13, respectively).
Intensity of experienced adverse events | 24 hours, 14 days and 28 days after each treatment administration
  Intensity of the experienced adverse events will be measured on a 11-point Numerical Rating Scale (e.g., "To what extent have you been feeling fatigue/dizziness?"; 0=not at all; 10=worst imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Lene Vase, MSc, PhD, DMSc, Principal Investigator — Dept. of Psychology and Behavioural Sciences, Aarhus University, Aarhus, Denmark
Locations (2):
- Denmark (2):
  - Department of Psychology and Behavioral sciences, Aarhus BSS, Aarhus University, Aarhus C, Denmark
  - Department of Clinical Medicine, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No